CLINICAL TRIAL: NCT02266329
Title: Chronic Postconcussive Headache: A Placebo-Controlled Treatment Trial of Prazosin
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: N1136-W; 1IK2RX001136-01A2 (NIH)
Record Dates: First submitted 2014-10-10; First posted 2014-10-17 (Estimated); Results first posted 2024-06-26 (Actual); Last update posted 2024-06-26 (Actual); Status verified 2024-06

CONDITIONS: Posttraumatic Headache; Combat Disorders; Post Concussion Syndrome; Headache; Mild Traumatic Brain Injury; Posttraumatic Migraine
Keywords: controlled clinical trial; randomized controlled clinical trial
MeSH Terms: conditions — Post-Traumatic Headache; Combat Disorders; Post-Concussion Syndrome; Headache; Brain Concussion | interventions — Prazosin

STUDY DESIGN:
Intervention Model Description: Randomized double blind placebo-controlled clinical trial with 2:1 chance of randomization to active drug.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- prazosin (Active Comparator): Subjects will be gradually titrated up to the maximum dose or the maximum tolerated dose based on a dosing algorithm. The maximum dose to be used in this trial is 5mg in the morning and 20 mg at bedtime.
  Interventions: Drug: prazosin hydrochloride
- placebo (Placebo Comparator): Subjects will be gradually titrated up to the maximum dose or the maximum tolerated dose based on a dosing algorithm. The maximum dose to be used in this trial is 5mg in the morning and 20 mg at bedtime.
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: prazosin hydrochloride — Prazosin as oral capsules titrated to the maximum dose or the maximum tolerated dose based on a dosing algorithm. The maximum dose to be used in this trial is 5mg in the morning and 20 mg at bedtime.
  Other Names: Minipress
  Arms: prazosin
Drug: placebo — Oral capsules of placebo identical in appearance to prazosin capsules titrated in the same manner as prazosin.
  Other Names: inactive drug; sugar pill; dummy pill
  Arms: placebo

SUMMARY:
The purpose of this study is to determine if prazosin is more effective than placebo in decreasing frequency, severity, disability, and other negative effects of headaches related to mild traumatic brain injury in Service Members and Veterans.

DETAILED DESCRIPTION:
Headaches following combat-related post-concussive injury are common, and in some patients can increase in frequency and severity to become very debilitating. Posttraumatic headaches (PTHAs), particularly those following blast-related head injury, can be resistant to standard headache therapies. The objective of this study is to evaluate the effectiveness of the medication prazosin as a prophylactic (preventive) agent in treating combat-related PTHAs. Prazosin is a generic drug originally marketed over 30 years ago as a treatment for high blood pressure. It has subsequently been found to be safe and effective for treating other problems, including most recently posttraumatic stress disorder (PTSD) and disrupted sleep in active duty Iraq/Afghanistan Service Members and Veterans. In preliminary studies, prazosin has also been found to substantially reduce the intensity and frequency of PTHAs in this population. This finding is the motivation behind this study.

The investigators' hypotheses are (1) that prazosin will be more effective than placebo in easing the effects of chronic PTHAs, including headache frequency, duration, severity, use of abortive/analgesic medications, and disability caused, and (2) that improvement in headache parameters will be associated with improvement in sleep quality, PTSD symptom severity, mood, cognition, health-related quality of life, and global clinical status, and with moderation of alcohol consumption.

The total trial length is 22 - 24 weeks. Following an initial clinic visit to determine preliminary study eligibility, there will be a 4-week pre-treatment preliminary screening period, during which participants will keep a daily headache diary. The purpose of this is to confirm eligibility for randomization per inclusion/exclusion criteria and to collect baseline data for headache-related outcome measures. Participants confirmed to be eligible to continue in the study will then have a one-week sleep evaluation including actigraphy and keeping a daily sleep diary. This will be followed by a baseline study visit, during which baseline data for secondary outcome measures will be collected using validated structured self-reports and clinician interviews. Participants will be randomized 2:1 to prazosin or placebo, and the study drug dose will be gradually titrated over a 5 to 7-week period to 5 mg in the morning and 20 mg in the evening or the maximum tolerated dose. The dose titration will be followed by 12 weeks at steady-dose. For the last week of the steady-dose phase, participants will repeat the sleep evaluation. Participants will keep a headache log through the duration of the study. Results will be analyzed using standard statistical techniques.

ELIGIBILITY:
Inclusion Criteria:

* Veterans or active duty service members aged 18 or older of either gender
* Good general health
* History of blast and/or impact head/neck trauma meeting DVBIC criteria for mild TBI, i.e., injury as manifested by at least one of the following:

  * 1) any period of loss of consciousness
  * 2) any loss of memory for events immediately before or after the accident
  * 3) any alteration in mental status at the time of the accident (e.g., feeling dazed, disoriented, or confused)
  * 4) focal neurological deficit(s) that may or may not be transient, with severity of injury not exceeding loss of consciousness 30 minutes, Glasgow Coma Scale <13-15 after 30 minutes, or posttraumatic amnesia >24 hrs,
* Headaches that started within 3 months of a head/neck injury or pre-existing headaches that markedly worsened (by a two-fold or greater increase in frequency and/or severity) within 3 months of a head/neck injury. Headaches must either 1) last 4 or more hours a day and reach a moderate to severe intensity at any point during the headache or 2) may be of any severity or duration if the participant uses a medication or other agent in an effort to stop the headache. Headaches meeting these criteria must have been present on average at least 8 days per 4-week period over the 3 months preceding study enrollment.
* Comorbid PTSD or other anxiety disorder is not exclusionary.
* Fluency in English is required.
* Persons of all races and ethnicities are eligible.
* Female participants must agree to abstain from sexual relations that could result in pregnancy or use a reliable form of birth control during the study.
* Continued use of prophylactic migraine medication other than the study drug is permissible if the participant has been on a stable dose for at least 4 weeks prior to the preliminary screening period and intends to continue the medication for the duration of the trial.

Exclusion Criteria:

* Participation in other interventional research.
* History of TBI more severe than that classified as mild by DVBIC criteria
* A primary non migraine and/or tension-type headache disorder that accounts for the majority of current symptoms
* History of penetrating head injury
* Headaches of any kind of moderate or severe intensity on an average of more than 4 days per month preceding the concussive trauma
* Acute or unstable chronic medical illness (e.g., unstable angina, myocardial infarction within 6 months, congestive heart failure, symptomatic or concerning cardiac arrhythmias; pre-existing hypotension (systolic BP<110) or orthostatic hypotension (systolic drop >20 mm mercury (Hg) after 2 min standing accompanied by lightheadedness). Also exclusionary are chronic renal or hepatic failure, Meniere's disease, insulin-dependent diabetes, diagnosed but untreated sleep apnea, history of epilepsy, stroke, dementia, active psychosis or psychotic disorder, severe depression, severe psychiatric instability or severe situational life crises, including evidence of being actively suicidal or homicidal, dementia, delirium within the prior 3 months. Other conditions will be evaluated on a case-by-case basis.
* Current substance use disorder per DSM-V criteria except caffeine- or tobacco-related disorders.
* Structural brain abnormalities on any prior imaging with associated clinically evident manifestations.
* Current participation in transcranial magnetic stimulation studies.
* Unable to reliably keep the headache log on a minimum of 80% of recordable days
* Women of childbearing potential must not be pregnant, planning to become pregnant during the study period, or nursing.
* Participation in a headache support group or other activity such as meditation or yoga intended to mitigate headache or other chronic pain must be stable for at least 4 weeks prior to beginning the preliminary screening period and should be intended to be continued for the duration of the trial. Participants will be encouraged to defer enrolling in such activities until they have completed the treatment trial.

Medication Exclusions:

Please note that the following two exclusions related to prazosin use had been changed in the study protocol as of September 2021 but were inadvertently not updated on the ClinicalTrials.gov website. The previous exclusion related to prazosin use prior to study enrollment was for a dose up to 2 mg. The change allows a dose up to 4 mg. This change, made based on clinical experience for the purpose of facilitating recruitment, did not adversely affect patient safety or data integrity.

* Past use of prazosin at a dose >4 mg is exclusionary.
* Current use of prazosin at a dose of 4 mg or less is not excluded, however requires a 2-week wash-out period prior to beginning the baseline headache log-keeping period.
* Current use of an alpha-1 antagonist for any purpose is exclusionary unless discontinued for at least 2 weeks prior to study entry and for the duration of a participant's study enrollment.
* Allergy or previous adverse reaction to prazosin or other alpha-1 antagonist
* Subjects must be on a stable dose of the following medications/treatments for at least 4 weeks prior to the preliminary screening period, and must intend to continue the medication for the duration of the trial: psychoactive drugs, for example anticonvulsants, benzodiazepines, antidepressants, sedative/hypnotics; antihypertensive medications, including beta blockers, calcium channel blockers, angiotensin converting enzyme inhibitors, and angiotensin receptor blockers; magnesium prescribed specifically for headache.
* Potential participants who have been taking trazodone will undergo a 2-week washout period before beginning the preliminary screening period. Because combining prazosin and trazodone may increase risk of priapism, trazodone is not allowed during the study.
* Sildenafil (Viagra), tadalafil (Cialis), vardenafil (Levitra), and avanafil (Stendra) will not be permitted during the dose titration period, because of increased risk of hypotension in combination with alpha-1 blockers, but will be allowed at half the usual starting dose following the study drug dose titration period, per VA prescribing guidelines.
* Use of butalbital within 4 weeks of beginning the preliminary screening period through the end of study involvement.
* Use of supplements containing nitrates and supplements containing stimulants (such as ephedra) within 2 weeks of beginning the preliminary screening period through the end of study involvement.
* Use of prescribed stimulants (such as amphetamine or dextroamphetamine containing medications) within 2 weeks of beginning the preliminary screening period through the end of study involvement.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 89 (Actual)
Dates: Start 2016-01-04 (Actual); Primary Completion 2023-05-31 (Actual); Study Completion 2023-09-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Cynthia L Mayer, DO, Principal Investigator — VA Puget Sound Health Care System Seattle Division, Seattle, WA
Locations (1):
- VA Puget Sound Health Care System Seattle Division, Seattle, WA, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 166 participants completed the informed consent process, agreeing to participation. 77 of those participants failed the screening process, declined to participate prior to study drug randomization, or were lost to follow-up prior to study drug randomization. 89 participants were randomized to study drug.
Period: Overall Study
Arm/Group | Prazosin | Placebo
Started (Subjects Randomized) | 59 | 30
Completed | 52 | 26
Not Completed | 7 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Prazosin | Placebo | Total
Number analyzed (Participants) | 59 | 30 | 89
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 1 | 00 | 1
  Between 18 and 65 years | 57 | 30 | 87
  >=65 years | 1 | 0 | 1
Age, Continuous [Mean (Standard Deviation); unit: years] | 38.6 (11.9) | 37.6 (10.1) | 38.3 (11.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 5 | 11
  Male | 53 | 25 | 78
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 11 | 5 | 16
  Not Hispanic or Latino | 34 | 20 | 54
  Unknown or Not Reported | 14 | 5 | 19
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaskan Native | 2 | 0 | 2
  Asian | 2 | 1 | 3
  Black | 12 | 8 | 20
  White | 31 | 18 | 49
  Hawaiian Native or Pacific Islander | 2 | 0 | 2
  Missing/Unknown | 3 | 0 | 3
  More than one race | 5 | 0 | 5
  Other | 2 | 3 | 5
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 59 | 30 | 89
Headache frequency [Mean (Standard Deviation); unit: headaches] — Number of headaches in the 4 weeks preceding baseline
  headaches | 15.5 (6.1) | 17.1 (6.0) | 16.0 (6.1)

OUTCOME MEASURES:

1. Primary Outcome: Headache Diary
Description: Change from baseline (pre-treatment) to Week 12 (i.e., following 12 weeks of drug treatment) of either 1) Headaches that last 4 or more hours a day and reach a moderate to severe intensity at any point or 2) Headaches of any intensity if a medication or other treatment is used in an effort to stop the Headaches, as determined from Headache Log data.
Time Frame: Baseline to 12 weeks
Measure: Mean (Standard Error); unit: headaches per month
Arm/Group | Prazosin | Placebo
Number analyzed (Participants) | 59 | 30
headaches per month | -10.7 (0.9) | -6.9 (1.3)
Statistical Analysis 1: Comparison: Prazosin vs Placebo; Change from baseline in headache (HA) frequency (1. Primary Outcome Measure) is based on linear mixed effects regression of outcome on study visit by treatment interaction with study participant as a random effect; Test type: Superiority; p = 0.034, Mixed Models Analysis — The significance of the study visit by treatment interaction with study visit coded as baseline, 4 weeks, 8 weeks, and 12 weeks; Mean Difference (Net) = -3.9, 95% CI 2-sided [-6.9 to -0.8], Standard Error of Mean 1.6

2. Secondary Outcome: Change From Baseline in 4-week Average Peak HA Severity
Description: Change from baseline (pre-treatment) to Week 12 (i.e., following 12 weeks of drug treatment) in 4-week average peak HA severity, as determined from Headache Log data.
Time Frame: Baseline to 12 weeks
Reporting Status: Not Posted

3. Secondary Outcome: Change From Baseline in 4-week Average Total Number of Hours of HA Pain
Description: Change from baseline (pre-treatment) to Week 12 (i.e., following 12 weeks of drug treatment) in 4-week average total number of hours of HA pain of any severity, as determined from Headache Log data.
Time Frame: Baseline to 12 weeks
Reporting Status: Not Posted

4. Secondary Outcome: Change From Baseline in Frequency of Use of Abortive/Analgesic Agents
Description: Change from baseline (pre-treatment) to Week 12 (i.e., following 12 weeks of drug treatment) in 4-week average frequency of use of abortive and/or analgesic HA treatment medications, as determined from Headache Log data.
Time Frame: Baseline to 12 weeks
Reporting Status: Not Posted

5. Secondary Outcome: Change From Baseline in Headache-Related Disability
Description: Change from baseline (pre-treatment) in average headache-related disability, as measured 1) in 4-week treatment intervals using the Headache Impact Test-6 and 2) in the full 12-week treatment interval using the Migraine Disability Assessment (for subjects who meet diagnostic criteria for migraine).
Time Frame: Baseline to 12 weeks
Reporting Status: Not Posted

6. Secondary Outcome: Change From Baseline in Posttraumatic Stress Disorder (PTSD) Symptoms
Description: Change from baseline (pre-treatment) in PTSD symptom severity, as measured using the PTSD Checklist (PCL) given at baseline and at 4-week treatment intervals.
Time Frame: Baseline to 12 weeks
Reporting Status: Not Posted

7. Secondary Outcome: Change From Baseline in Sleep Measures
Description: Change from baseline (pretreatment) in sleep characteristics, including sleep quality, quantity, and efficiency using 1) the Pittsburgh Sleep Quality Index and the Insomnia Severity Index given at baseline and at 4-week treatment intervals and 2) sleep diary and wrist actigraphy performed for one week at baseline and after 11 weeks of treatment
Time Frame: Baseline to 12 weeks
Reporting Status: Not Posted

8. Secondary Outcome: Change From Baseline in Concussion-Related Symptoms
Description: Change from baseline (pre-treatment) in concussion-related symptoms, as measured at 4-week treatment intervals using the Neurobehavioral Symptom Inventory
Time Frame: Baseline to 12 weeks
Reporting Status: Not Posted

9. Secondary Outcome: Change From Baseline in Depressive Symptoms
Description: Change from baseline (pre-treatment) in depressive symptoms, as measured at 4-week treatment intervals using the Patient Health Questionnaire-9.
Time Frame: Baseline to 12 weeks
Reporting Status: Not Posted

10. Secondary Outcome: Change From Baseline in Alcohol Use
Description: Change from baseline (pre-treatment) in alcohol use, as measured at 4-week treatment intervals using the Alcohol Use Disorders Identification Test-Consumption.
Time Frame: Baseline to 12 weeks
Reporting Status: Not Posted

11. Secondary Outcome: Change From Baseline in Global Cognitive Function
Description: Change from baseline (pre-treatment) in cognitive function, as measured at 4-week treatment intervals using the Montreal Cognitive Assessment (MoCA).
Time Frame: Baseline to 12 weeks
Reporting Status: Not Posted

12. Secondary Outcome: Change From Baseline in Pupillary Light Responses
Description: Change from baseline (pre-treatment) to Week 12 (i.e., following 12 weeks of drug treatment) in pupillary light responses using pupillometry, as a measure of sympathetic activation.
Time Frame: Baseline to 12 weeks
Reporting Status: Not Posted

13. Secondary Outcome: Photophobia
Description: Change from baseline (pre-treatment) to Week 12 (i.e., following 12 weeks of drug treatment) in light sensitivity symptoms, as determined using a modified Utah Photophobia Symptom Impact Scale - 12-Item)
Time Frame: Baseline to 12 weeks
Reporting Status: Not Posted

14. Secondary Outcome: Number of Patients With a 50% or More Decrease in Mean Number of Headache Days Per 4 Weeks
Description: Number of patients with a 50% or more decrease in mean number of headache days per 4 weeks, as determined at 4 week treatment intervals using Headache Log data.
Time Frame: Baseline to 12 weeks
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 24 weeks
Arm/Group | Prazosin | Placebo
All-Cause Mortality (participants affected / at risk) | 0/59 | 0/30
Serious Adverse Events (participants affected / at risk) | 1/59 | 1/30
Other Adverse Events (participants affected / at risk) | 52/59 | 22/30
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Prazosin (N=59) | Placebo (N=30)
Planned surgical procedure (Surgical and medical procedures) | 1 (1) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Prazosin (N=59) | Placebo (N=30)
Palpitations (Cardiac disorders) | 21 (23) | 6 (6)
Nausea (Gastrointestinal disorders) | 20 (25) | 4 (4)
Dizziness (any) (General disorders) | 37 (51) | 6 (7)
Dizziness on Standing (General disorders) | 24 (30) | 1 (1)
Drowsiness/Lethargy (General disorders) | 26 (30) | 5 (5)
Insomnia (General disorders) | 8 (10) | 2 (2)
Lightheadedness (General disorders) | 28 (32) | 11 (11)
Low Energy (General disorders) | 16 (17) | 3 (3)
Nasal Congestion (General disorders) | 19 (21) | 3 (3)
Peripheral Edemna (General disorders) | 11 (12) | 3 (4)
Vertigo (General disorders) | 1 (1) | 1 (1)
Weakness (generalized) (General disorders) | 6 (6) | 1 (1)
Headache worsening (General disorders) | 2 (2) | 4 (5)
Depression or depressed mood (Psychiatric disorders) | 7 (7) | 2 (2)
Suicidal Ideation (Psychiatric disorders) | 3 (3) | 0 (0)
Incontinence (Renal and urinary disorders) | 4 (4) | 0 (0)

LIMITATIONS AND CAVEATS:
Change from baseline in headache (HA) frequency (1. Primary Outcome Measure) is based on linear mixed effects regression of outcome on study visit by treatment interaction with study participant as a random effect.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-11-12): https://cdn.clinicaltrials.gov/large-docs/29/NCT02266329/Prot_SAP_000.pdf